CLINICAL TRIAL: NCT02175251
Title: Low and High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Resistant Auditory Hallucination in Schizophrenia: a Double Blind Sham-controlled Randomised Study
Brief Title: Low and High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Resistant Auditory Hallucination in Schizophrenia
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P120909; IDRCB 2013-A00872-43 (Other: FRENCH AUTHORITY)
Record Dates: First submitted 2014-05-22; First posted 2014-06-26 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia
Keywords: rTMS; Schizophrenia; high frequency rTMS; low frequency rTMS; AHRS; SAPS SANS PANSS; GAF; UKU
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low frequency (1Hz) (Active Comparator): low frequency
  Interventions: Procedure: low frequency (1Hz)
- Sham Comparator (Sham Comparator): Sham Comparator
  Interventions: Procedure: Sham Comparator
- high frequency (20Hz) (Experimental): high frequency
  Interventions: Procedure: high frequency (20Hz)

INTERVENTIONS:
Procedure: high frequency (20Hz) — 10 session in 5 days with high frequency (20 Hz)
  Arms: high frequency (20Hz)
Procedure: low frequency (1Hz) — 10 session in 5 days with low frequency (1Hz)
  Arms: low frequency (1Hz)
Procedure: Sham Comparator — 10 session in 5 days with sham-controlled
  Arms: Sham Comparator

SUMMARY:
Auditory Hallucinations (AH) are experienced by 50 to 70% of subjects with schizophrenia. Almost a quarter of patients are medication resistant to such symptoms. The application of rTMS at low frequency in the left temporoparietal cortex reduces AH. A pilot study reported successful treatment of AH with high frequency rTMS. rTMS (20Hz) should be a shorter and an easier treatment for out-patients with schizophrenia compared to low stimulation treatment.

DETAILED DESCRIPTION:
90 schizophrenia patients Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM IV-TR) criteria with persistent Auditory Hallucinations (AH) resistant to antipsychotic treatments will be recruited. A double blind sham-controlled randomized parallel study comparing three groups treated 10 session in 5 days with high frequency (20 Hz), low frequency (1Hz) and sham-controlled condition rTMS. They will be followed 3 month and evaluated using Auditive Hallucination Rating Scale (AHRS), Scale for the Assessment of Positive Symptoms Scores (SAPS), Scale for the Assessment of Negative Symptoms Scores (SANS) and Positive And Negative Symptom Scale (PANSS) global score and Global Assessment of Functioning (GAF) score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia DSM IV-TR criteria and persistent AH resistant to antipsychotic treatments.

Exclusion Criteria:

* Left handed patients lateralizes
* rTMS contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2017-07-07 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficiency of high frequency (20Hz) repetitive Transcranial Magnetic Stimulation (rTMS) to the left temporoparietal cortex compared to sham controlled condition rTMS in term on Auditory Hallucinations reduction. | 5 day
  Auditory Hallucinations improvement at 5-day was evaluate with AHRS (Auditory Hallucination Rating Scale) score

SECONDARY OUTCOMES:
To compare the efficiency of low frequency (1Hz) to sham-controlled condition repetitive Transcranial Magnetic Stimulation (rTMS) in term of Auditory Hallucination reduction. | 5 days
  Auditory Hallucinations improvement evaluated with Auditory Hallucination Rating Scale (AHRS)
To compare the efficiency of high frequency to low frequency (1Hz) in term of Auditory Hallucination reduction. | 5 days
  Auditory Hallucinations improvement evaluated with Auditory Hallucination Rating Scale (AHRS)
To compare the maintenance of therapeutic effect for one month of high frequency to low frequency (1Hz) in term of Auditory Hallucination reduction. | 1 month
  Auditory Hallucinations improvement evaluated with Auditory Hallucination Rating Scale (AHRS)
To evaluate the maintenance of therapeutic effect of high frequency compared to sham controlled condition for 15 days 1 month, 2 months and 3 months | 15 days 1 month, 2 months and 3 months
To compare the side effects of each of the active treatment | at Inclusion and 5 day
  Tolerance assessed with the UDVALG of KLINISKE UNDERSOGELSER scale (UKU )

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DUBERTRET, PU-PH, Study Director — Department of Psychiatry, Louis MOURIER Hospital
Locations (1):
- Department of Psychiatry, Louis Mourier Hospital, Colombes, France